CLINICAL TRIAL: NCT03975803
Title: Reliability and Responsiveness of the Chinese Version of the Readiness for Return-To-Work Scale in Lost-time Claimants in Outpatient Occupational Rehabilitation in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201904067RINC
Record Dates: First submitted 2019-06-02; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Occupational Injuries
Keywords: return to work; readiness for return to work; occupational injury; work hardening
MeSH Terms: conditions — Occupational Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to measure the reliability and responsiveness of the Chinese version of the readiness for return-to-work (RRTW) scale. We would conduct a multiple-centered, prospective cohort study to require RRTW data in lost-time claimants in outpatient occupational rehabilitation in Taiwan.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of occupational injuries
* Participating the work hardening program
* Age from 20-65
* Still not return to work
* Willing to participating the study

Exclusion criteria:

* Cannot read the sentences or express their own idea, which causing the cannot finish the questionnaires
* Brain injuries (e.g. traumatic brain injury, cerebrovascular acciden

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 lost-time claimants in outpatient occupational rehabilitation in 3 work hardening centers in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-03 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of the Readiness for Return-To-Work Scale scores during rehabilitation | The participants do the pretest of RRTW scale in the first week in their work hardening program, finishing the protest in the last week before the program ends. The duration depends on people. (In an average of 4-6 weeks)
  Using the RRTW scale changes of the pretest and protest data to calculate the responsiveness.

SECONDARY OUTCOMES:
Change from the Readiness for Return-To-Work Scale scores at 1 week | The participants do the pretest of RRTW scale in the first week in their work hardening program, and they do the retest after one week.
  Using the pretest and retest data of the Readiness for Return-To-Work (RRTW) scale to calculate the reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Keh-Chung Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan